CLINICAL TRIAL: NCT05175027
Title: "Comparison of Povidone Iodine and Hypochlorous Acid Used as a Preoperative Antiseptic in Neonatal Circumcision"
Brief Title: Preoperative Antiseptic in Newborn Circumcision Comparison of Povidone Iodine and Hypochlorous Acid Used
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hisar Intercontinental Hospital (Other)
Responsible Party: Principal Investigator, Basri Cakiroglu, Ass. Prof., Hisar Intercontinental Hospital
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 2021/15
Record Dates: First submitted 2021-11-11; First posted 2022-01-03 (Actual); Last update posted 2022-01-03 (Actual); Status verified 2021-12

CONDITIONS: Newborn; Infection; Disinfection; Circumcision
Keywords: circumcision,; wound; antibacterial
MeSH Terms: conditions — Infections; Wounds and Injuries | interventions — Hypochlorous Acid; Povidone-Iodine

STUDY DESIGN:
Intervention Model Description: Two models:Newborns to be circumcised randomly were divided into two groups as Hypochlorosis group and Povidone iodine group.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypochlorosis (Active Comparator): Hypochlorosis was used as an antiseptic for the patients
  Interventions: Drug: hypochlorous acid
- Povidone iodine (Active Comparator): Povidone iodine was used as an antiseptic for the patients
  Interventions: Drug: hypochlorous acid

INTERVENTIONS:
Drug: hypochlorous acid — Randomize
  Other Names: povidone iodine

SUMMARY:
Comparison of Povidone iodine and Hypochlorous acid used as a Preoperative Antiseptic in Newborn Circumcision abstract

Aim:

Circumcision is one of the most common surgical procedures in all age groups. Before the circumcision procedure, asepsis is provided with a surface disinfectant. Various methods can be used for this process. Povidone iodine, which has been used for years during the transition from traditional circumcision methods to surgical circumcision methods; tissue damage, allergic reactions and increase in pain level. For this reason, the investigators aimed to compare it with Hypochlorous acid (Crystalin), which is a less toxic and more physiological antiseptic solution.

Material and Method:

Newborns to be circumcised randomly were divided into two groups as Hypochlorosis group and Povidone iodine group. At the beginning of the circumcision procedure, a culture was taken in the form of a prepucial swab 1 minute after the cleaning of the local area and the inner surface of the prepuce. Then circumcision was performed. Culture results and complications were compared.

DETAILED DESCRIPTION:
It is aimed to compare two solutions used for cleaning the operation area in newborn circumcision.It was conducted to compare the antibacterial activity of povidone iodine and hypochlorous.

ELIGIBILITY:
Inclusion Criteria:

* male
* newborn,

Exclusion Criteria:

* hipospadias,
* epispadias,
* urinary infectious

Ages: 1 Day to 1 Month | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — male
Enrollment: 60 (Actual)
Dates: Start 2021-05-05 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2021-11-11 (Actual)

PRIMARY OUTCOMES:
The effect of both drugs on wound healing will be investigated. | one month
  there is wound healing;1,no wound healing:0
The effect of both drugs on antibacterial effects will be investigated | one week
  there is bacterial growth:1, there is no bacterial growth:0

CONTACTS AND LOCATIONS:
Overall Officials: Basri Cakiroglu, Study Director — Hisar Intercontinental Hospital
Locations (1):
- Hisar Intercontinental Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No